CLINICAL TRIAL: NCT02631252
Title: A Phase I Study of Combination Chemotherapy With Mitoxantrone and Etoposide (VP-16) Combined With an Autophagy Inhibitor, Hydroxychloroquine (HCQ), for the Treatment of Patients With Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: Phase I Study of Mitoxantrone and Etoposide Combined With Hydroxychloroquine, for Relapsed Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to accrue
Sponsor: Alison Sehgal, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Alison Sehgal, MD, MS, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-133
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Leukemia, Acute Myelogenous
Keywords: Leukemia; Acute Myelogenous; Phase I; Mitoxantrone; Etoposide; Hydroxychloroquine; Relapsed; Autophagy inhibitor; AML; Relapsed AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Recurrence | interventions — Hydroxychloroquine; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label, Single-arm (Experimental): Hydroxychloroquine + Mitoxantrone + Etoposide
  Hydroxychloroquine is given up to 21 days, started concurrently with both Mitoxantrone, administered by IVPB over 15 minutes each day for 5 days and Etoposide, administered intravenously over 2 hours each day for 5 days
  Interventions: Drug: Hydroxychloroquine; Drug: Mitoxantrone; Drug: Etoposide

INTERVENTIONS:
Drug: Hydroxychloroquine — Doses ranging from 600-1400mg daily in divided twice daily doses and administered orally.
  Other Names: Plaquenil
Drug: Mitoxantrone — Dose: 10mg/m2 IVPB in 50ml NS
  Other Names: Dihydroxyanthracenedione, DHAD
Drug: Etoposide — Dose: 100 mg/m2 administered intravenously in 500 ml of 0.9% sodium chloride
  Other Names: Toposar®; EPEG

SUMMARY:
This is an open label phase I clinical trial of hydroxychloroquine (HCQ) ,when it is combined with the usual medications for acute myeloid leukemia, mitoxantrone and etoposide. The purpose of this study is to find the safest and most effective dose of hydroxychloroquine with these medications. The investigators will be testing to see if it can increase the effectiveness of mitoxantrone and etoposide.

DETAILED DESCRIPTION:
Hydroxychloroquine is not FDA (United States Food and Drug Administration) approved for AML and is considered an investigational drug in this study. It has helped make chemotherapy more effective in animals. The investigators will be testing to see if it can increase the effectiveness of mitoxantrone and etoposide. It has been combined with other types of chemotherapy for humans with other types of cancer. Most of the patients were able to take hydroxychloroquine safely at the doses studied in this clinical trial.

Hydroxychloroquine is approved by the FDA for malaria, rheumatoid arthritis, and other autoimmune diseases. Mitoxantrone is approved by the FDA for use in AML, and it is one of the most common drugs used in the treatment of AML. Etoposide is not approved by the FDA for AML. It is approved for small cell lung cancer and testicular cancer. It is commonly used in AML.

The primary objective of this trial is to determine the recommend phase 2 dose (RP2D) for HCQ combined with mitoxantrone and etoposide, while secondary objectives include efficacy estimates of this combination at the RP2D, a safety and tolerability profile of this combination, as well as the correlation of pharmacodynamic assessments of autophagy inhibition with dose and clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and have the ability to provide written consent
2. Age > 18 years old to <80 years old
3. Patients with AML in the first morphologic relapse as defined by >5% reappearance of leukemia blasts in the bone marrow not attributable to any other cause (Appendix I) who have not yet received chemotherapy for the current relapse
4. Eastern Cooperative Oncology Group Performance Status of 0 -2 (see Appendix II)
5. Adequate organ function

   1. Serum creatinine ≤ 1.5 mg/dl and calculated creatinine clearance ≥ 50 mL/min (using the Cockcroft-Gault equation CL creatinine = (140-age) x body mass X 0.85 if female)/72 x creatinine where age is given in years, body mass is given in kg and creatinine is given in mg/dL)
   2. Aspartate aminotransferase (AST) ≤ 5x the upper limit of normal Alanine aminotransferase (ALT) < 5x the upper limit of normal
   3. Direct bilirubin ≤ 1.5 mg/dl Note: As many eligible patients will be pancytopenic secondary to their disease or prior treatments, hematologic abnormalities will not be used as a criteria for entry or exclusion
6. Left ventricular ejection fraction (LVEF) ≥50 %
7. Females of child-bearing potential must have a negative pregnancy test during screening and all subjects must agree to use an effective method of contraception. A woman is eligible to enter and participate in the study if she is of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who has had a hysterectomy or has had a bilateral oophorectomy (ovariectomy).
   2. Childbearing potential, has a negative serum pregnancy test during the screening period and agrees to avoid sexual activity or use accepted methods of contraception from screening through follow-up.

Men with a female partner of childbearing potential are eligible to enroll and participate in the study if they have had either a prior vasectomy or agree to avoid sexual activity or use appropriate barrier contraception from screening through post-treatment follow-up.

Exclusion Criteria:

1. Acute promyelocytic leukemia
2. Prior chemotherapy regimen given for 1st relapse, not including the use of hydroxyurea or plasmapheresis that is used prior to the initiation of chemotherapy.
3. Previous use of mitoxantrone and etoposide combination therapy within the preceding 180 days of screening.
4. Symptomatic central nervous system (CNS) involvement
5. Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
6. History of psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
7. Current receiving any other anti neoplastic investigational agents
8. Prior autologous or allogeneic stem cell transplantation
9. Concurrent malignancy. Exceptions: Patients who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with concurrent malignancies that are indolent or definitely treated may be enrolled.
10. Women who are pregnant or breastfeeding
11. Evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory or cardiac disease)
12. Inability to take oral medications, due to impaired swallowing ability or poor absorption capacity
13. Known glucose-6-phosphate dehydrogenase (G-6PD) deficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2016-09-17 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Select a recommended phase 2 dose (RP2D) for hydroxychloroquine | during the first 7 weeks after initiating therapy
  Dose limiting toxicity (DLT) that occurs during the first 7 weeks after initiating therapy and is at least possibly related

SECONDARY OUTCOMES:
Complete Remission (CR) | up to 4 weeks after completion of therapy
Overall Survival (OS) | until death or last patient contact, up to 5 years
Relapse Free Survival (RFS) | until relapse or death, whichever occurs first, or last patient contact, for up to 5 years
Pharmacodynamic Endpoint - Measurement of LC3-1 | up to 4 weeks after completion of therapy
Pharmacodynamic Endpoint - Measurement of LC3-2 | up to 4 weeks after completion of therapy
Pharmacodynamic Endpoint - Measurement of p62 | up to 4 weeks after completion of therapy
Pharmacodynamic Endpoint - Measurement of HMGB1 | up to 4 weeks after completion of therapy
Pharmacodynamic Endpoint - Measurement of RAGE | up to 4 weeks after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alison Sehgal, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute - Hillman Cancer Center, Pittsburgh, Pennsylvania, United States